CLINICAL TRIAL: NCT05684718
Title: A Phase 1 Single Center Open-label, Non-randomized, Fixed Sequence Study in Healthy Volunteers to Assess the Pharmacokinetics (PK) of BV100 When Administered Alone and With Itraconazole
Brief Title: To Evaluate the Effect of Multiple Doses of Itraconazole on the Pharmacokinetics of BV100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Collaborators: Clinical Research Units Hungary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV100-007
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-01

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Rifabutin; Itraconazole

STUDY DESIGN:
Intervention Model Description: Fixed sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BV100 Plus Itraconazole (Experimental): A total 2 doses of BV100 and 14 doses of itraconazole will be administered to each participant per specified dosing schedule
  Interventions: Drug: BV100 (300 mg); Drug: Itraconazole 200 mg

INTERVENTIONS:
Drug: BV100 (300 mg) — Intravenous solution
  Other Names: Rifabutin for Infusion
Drug: Itraconazole 200 mg — Oral solution
  Other Names: Sporanox Oral solution

SUMMARY:
Phase I clinical study to evaluate the effect of multiple doses of itraconazole on the pharmacokinetics of BV100 in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence Phase I clinical study to evaluate the effect of multiple doses of itraconazole on the pharmacokinetics of rifabutin, 25 O deacetyl-rifabutin and DMI in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were able to understand and follow instructions during the study.
2. Subjects who signed informed consent.
3. Male subjects ≥18 and ≤55 years of age; female subjects ≥18 and ≤50 years of age of non-childbearing potential defined as follows:

   * Female subjects 50 years of age, in menopause for 24 consecutive months and not receiving any hormone replacement therapy within 24 months prior to inclusion into the study
   * Female subjects who underwent surgical sterilization
   * Female subjects who underwent hysterectomy
   * Female subjects with documented premature ovarian failure
4. Weight within a BMI range of 19.0-30.0 kg/m2.
5. Estimated glomerular filtration rate (eGFR) according to the CKD-EPI: ≥90 mL/min (normal renal function)
6. Healthy subjects have to be in a good health in the opinion of the study physician, as determined by medical history, ECG, vital signs, physical examination, and clinical laboratory tests.
7. Having had no febrile or infectious illness for at least 14 days prior to dosing.
8. The subject was available to complete the study.
9. The subject is willing to comply with the restrictions and requirements of the protocol and, in the opinion of the study physician, will be able to complete the study.

Exclusion Criteria:

1. Unwilling or unable to give informed consent.
2. As a result of the medical screening process, the study physician considered the subject unfit for the study.
3. Pregnant or lactating women or men with female partners who are lactating or are pregnant.
4. Known or suspected history of hypersensitivity to rifabutin or excipients or to drugs of a similar chemical class including rifampicin, rifapentine, rifaximin; history of allergic reactions leading to hospitalisation or any other allergic conditions (including drug allergies, asthma, eczema, anaphylactic reactions but excluding untreated, asymptomatic, seasonal allergies) which the Investigator considers may affect the safety of the subject and/or out-come of the study.
5. History of antibiotic associated diarrhoea within the last year.
6. Subjects with ECG abnormalities (history, or evidence of second-degree heart block of Mobitz type II, third degree heart block, or any abnormality considered relevant by the Investigator), QTcF > 450 ms, PR > 210 ms, or QRS duration > 115 ms.
7. Average supine systolic blood pressure > 140 mmHg or < 90 mmHg or average diastolic blood pressure > 90 mmHg or < 50 mmHg at Screening or Day 1 prior to dosing (any abnormal blood pressure results may be repeated once and if the repeat result is within the normal range, it is not considered to have met the exclusion criterion). Pulse rate > 90 or < 50 beats per minute at Screening or Day 1 prior to dosing.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and creatinine, above the ULN at Screening. Any abnormal value of these parameters may be repeated during screening period and if the repeat result is within the laboratory reference range, it is not considered to have met the exclusion criterion.
9. Screening values other than AST, ALT, ALP, creatinine, for haematology, biochemistry, or urinalysis must not exceed the reference range. Minor deviations from normal are allowed if they are not clinically significant.
10. History of symptomatic, chronic or recurrent infection (e.g. nausea, vomit-ing, diarrhoea, infection with fever) or any viral (including symptomatic herpes zoster), bacterial (including upper respiratory infection), fungal (non-cutaneous) or parasitic infection within 30 days prior to admission to the clinical unit.
11. A positive pre-study serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV)-1 and/or 2 antibodies.
12. Positive Coronavirus (SARS-CoV-2) rapid test and/or PCR (upon Check-in on Day -1). If a subject has negative rapid test but a positive PCR, the subject could be included if his/her medical history is consistent with pre-vious COVID-19 infection explaining his/her positive PCR within the last 90 days.
13. A positive pre-study drug/alcohol screen.
14. History of epilepsy, seizures, other neurological disorders, or neuropsychiatric conditions.
15. Subjects who have received any prescribed systemic or topical medication within 4 weeks of the first dose administration.
16. Subjects who had used any non-prescribed systemic or topical medication (including herbal remedies) or megadose vitamins (i.e. 20 to 600 times the recommended daily supplement dose) within 7 days prior to dosing, unless in the opinion of the study physician the medication did not interfere with the study procedures or compromise safety
17. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration.
18. Regular use of any inducer of metabolism (e.g., barbiturates, rifampin) in the3 months prior to the first dose administration.
19. Subjects who have participated in a clinical study involving administration of an investigational drug (new chemical entity) within the following time period prior to the first dose administration in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
20. Subjects who consume more than 21 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 30 mL of 40% of alcohol by volume distilled spirits).
21. Excessive consumption of caffeine- or xanthine-containing food or beverages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to study treatment administration.
22. Subjects who smoked more than 10 cigarettes a day.
23. Any use of drugs-of-abuse or alcohol abuse within 2 years prior to the first admission to the clinical unit.
24. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the requirements of the study.
25. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct. Failure to satisfy the Investigator of fit-ness to participate for any other reason.
26. Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.
27. Inability to refrain from using soft contact lenses starting from administration of study treatment until follow-up visit.
28. Subjects who are study site employees or immediate family members of the study site or Sponsor employee.
29. Contraindications related to itraconazole: decompensated heart failure, chronic obstructive pulmonary disease, concomitant administration of itraconazole and CYP3A4 metabolized drugs known to prolong the QT interval, may result in potentially fatal ventricular tachyarrhythmias, including torsades de pointe or a life-threatening arrhythmia. Hypersensitivity or previous adverse events associated with azole antifungals.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of repeated doses of itraconazole on the pharmacokinetics of intravenous rifabutin | Day 1 to Day 21
  maximum observed plasma concentration (Cmax) of rifabutin
To evaluate the effect of repeated doses of itraconazole on the pharmacokinetics of intravenous rifabutin | Day 1 to Day 21
  Area Under the Plasma Concentration-Time Curve (AUC) of rifabutin
To evaluate the effect of repeated doses of itraconazole on the pharmacokinetics of intravenous 25-O-deacetyl-rifabutin | Day 1 to Day 21
  maximum observed plasma concentration (Cmax) of 25-O-deacetyl-rifabutin
To evaluate the effect of repeated doses of itraconazole on the pharmacokinetics of intravenous 25-O-deacetyl-rifabutin | Day 1 to Day 21
  Area Under the Plasma Concentration-Time Curve (AUC) of 25-O-deacetyl-rifabutin

SECONDARY OUTCOMES:
Safety and tolerability of single doses of BV100 | 28 Days
  Number of Participants with Treatment -Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Husband, MD, Study Director — BioVersys SAS
Locations (1):
- CRU Hungary Kft., Early Phase Unit, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No